CLINICAL TRIAL: NCT05658822
Title: Enteric Dysmotility in Mitochondrial Neurogastrointestinal Encephalomyopathy Patients Detected by High-resolution
Brief Title: Digestive Dysmotility in Mitochondrial Neurogastrointestinal Encephalomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)56/2018E
Record Dates: First submitted 2022-11-27; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: MNGIE; Dysmotility
Keywords: Intestinal manometry; motility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mitochondrial neurogastrointestinal encephalopathy (MNGIE) is an ultra-rare mitochondrial disease caused by mutations of the gen that codifies the enzyme thymidine phosphorylase The genetic defect results in systemic accumulation of the nucleosides thymidine and deoxyuridine. Clinically MNGIE is characterized by a combination of gastrointestinal and neurological manifestations, including severe gastrointestinal dysmotility, cachexia, ptosis, external ophthalmoplegia and sensorimotor neuropathy. Gastrointestinal symptoms are the most frequent first manifestation of the disease, and include early satiety, nausea, dysphagia, postprandial emesis, abdominal pain, abdominal distention, and diarrhea. The disease is relentlessly progressive and the cause of death is primarily related to digestive dysmotility. However, the specific motor dysfunctions that produce the symptoms, i.e., the underlying mechanisms, remain uncertain.

DETAILED DESCRIPTION:
Mitochondrial neurogastrointestinal encephalopathy (MNGIE) is an ultra-rare mitochondrial disease caused by mutations of the gen that codifies the enzyme thymidine phosphorylase The genetic defect results in systemic accumulation of the nucleosides thymidine and deoxyuridine. Clinically MNGIE is characterized by a combination of gastrointestinal and neurological manifestations, including severe gastrointestinal dysmotility, cachexia, ptosis, external ophthalmoplegia and sensorimotor neuropathy. Gastrointestinal symptoms are the most frequent first manifestation of the disease, and include early satiety, nausea, dysphagia, postprandial emesis, abdominal pain, abdominal distention, and diarrhea. The disease is relentlessly progressive and the cause of death is primarily related to digestive dysmotility. However, the specific motor dysfunctions that produce the symptoms, i.e., the underlying mechanisms, remain uncertain, because so far, no studies on gastrointestinal motility in MNGIE have been published. The aims of this study were to identify the upper GI motor dysfunction in MNGIE patients, and to determine their relation to the clinical manifestations. Since the life-threatening consequences of the disease involve the upper gastrointestinal tract, all patients, after a thorough clinical and neurological evaluation, fulfilled a structured clinical questionnaire on digestive manifestations, and underwent state-of-the-art evaluation of the esophagus and the small bowel by high-resolution manometry (HRM), and gastric emptying by scintigraphy

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MNGIE disease established by thymidine phosphorylase activity and mitochondrial mutation analysis.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with MNGIE
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
intestinal motility at diagnosis | In patients included, in the first 30 days from diagnosis
  to assess the number of intestinal contractions (contractions per minute) during fasting and after the infusion of nutrients measured by high-resolution intestinal manometry
intestinal motility at diagnosis | In patients included, in the first 30 days from diagnosis
  to assess the amplitude (mmHg) of contractions during fasting and after nutrients measured by high-resolution intestinal manometry

SECONDARY OUTCOMES:
intestinal motility response to hepatic transplant | one and two years after hepatic transplant treatment
  to assess changes in the number of intestinal contractions (contractions per minute) during fasting and after the infusion of nutrients measured by high-resolution intestinal manometry after hepatic transplant
intestinal motility response to hepatic transplant | one and two years after hepatic transplant treatment
  to assess the amplitude of intestinal contractions during fasting and after the infusion of Amplitude (mmHg) of contractions during fasting and after nutrients measured by high-resolution intestinal manometry after hepatic transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No